CLINICAL TRIAL: NCT01411787
Title: Bootcamp During Neoadjuvant Chemotherapy for Breast Cancer "Can we Kick Down Ki-67, Punch Out Insulin Resistance, and Increase Survival?"
Brief Title: Bootcamp During Neoadjuvant Chemotherapy for Breast Cancer
Acronym: Bootcamp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 122010-150
Record Dates: First submitted 2011-08-02; First posted 2011-08-08 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer
Keywords: Breast cancer; neoadjuvant chemotherapy; exercise; Ki-67
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Patient will continue normal activities. Ki-67 will be measured in the initial core biopsy and then again in the final pathologic specimen which is removed for definitive surgical intervention. Insulin resistance levels will be measured by obtaining insulin-like growth factor binding protein one and C-peptide levels just prior to initiation of neoadjuvant chemotherapy, and then again after the last chemotherapy dose. Body mass index, percent body fat, and improving fitness levels will also be measured.
- Exercise (Experimental): Five woman undergoing neoadjuvant chemotherapy for breast cancer will be randomized to an exercise protocol supervised by an experienced personal trainer. The exercise will be administered three times a week for the 4-6 months of neoadjuvant chemotherapy. The exercise protocol will consist of activities including walking/running up to a mile, calisthenics, and light weightlifting.
  Ki-67 will be measured in the initial core biopsy specimen and then again in the final pathologic specimen which is removed for definitive surgical intervention. Insulin resistance levels will be measured by obtaining insulin-like growth factor binding protein one and C-peptide levels just prior to inititation of neoadjuvant chemotherapy and then again after the last chemotherapy dose in both arms. Body mass index, percent body fat, and improving fitness levels will also be measured.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Five woman undergoing neoadjuvant chemotherapy for breast cancer will be randomized to an exercise protocol supervised by an experienced personal trainer. The exercise will be administered three times a week for the 4-6 months of neoadjuvant chemotherapy. The exercise protocol will consist of activities including walking/running up to a mile, calisthenics, and light weightlifting.
  Arms: Exercise

SUMMARY:
This is a randomized, single-site pilot study incorporating one control group. This research involves an exercise group and a non-exercise group (control group).

The patients who are in the exercise group will be enrolled in the Dallas County Women's Adventure Boot Camp. This will require them to undergo exercise training 3 times per week, under the direction of an experienced personal trainer in a group setting. All Boot Camp personal trainers are trained in basic cardiac life support (CPR) and are trained to watch for any signs or symptoms associated with a poor exercise response.

The investigators hypothesize that randomizing women to a supervised exercise program of core conditioning, muscular/circuit training, and short distance running administered during neoadjuvant chemotherapy for breast cancer can be performed.

Patients will continue on study as they are undergoing neoadjuvant chemotherapy for their breast cancer. This will be about 4 - 6 months.

DETAILED DESCRIPTION:
The exercise protocol will consist of activities including walking/running up to a mile, calisthenics (jumping jacks, short relays, rapid punches) and light (no greater than 5 pounds) weight lifting. The patients who do not receive the exercise program will be allowed to do what they would normally do during their neoadjuvant chemotherapy. They are allowed to engage in their own exercise regimens and diet modifications.

Subjects will receive the chemotherapy as directed by their physicians, and then undergo surgery as planned. Randomization will occur by drawing cards entitled "exercise" or "control" from an envelope and then assigning the patient to this group.

ELIGIBILITY:
Inclusion Criteria:

1. Receiving neoadjuvant chemotherapy for breast cancer at one of the UT Southwestern hospitals or affiliates (Simmons Cancer Center, Parkland Hospital)
2. No evidence of metastatic disease as confirmed by routine staging
3. 18 - 70 year old female
4. Karnofsky score >80%
5. Body Mass Index >25 kg/m2
6. Able to speak, read and understand the English language
7. Ability to understand and willingness to sign a written informed consent document
8. All races and ethnicities will be eligible.

Exclusion Criteria:

1. Unable to speak, read and understand the English language
2. Patients may not be involved in other trials evaluating the efficacy of neoadjuvant therapy
3. Insulin-dependent diabetic patients.
4. Known to be pregnant or planning to become pregnant during the study.
5. Subjects are prohibited from being on other cancer treatments aside from what their treating medical oncologist has prescribed, primarily additional chemotherapies.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-03; Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
Ki-67 index | post-neoadjuvant chemotherapy; ~ 4-6 months from treatment start
  Ki-67 has significant value for predicting survival and recurrence risk in breast cancer. A recent study reveals that patients with a post-neoadjuvant chemotherapy Ki-67 index of less than 1.0% had significantly improved survivals when compared to patients with a Ki-67 index > 1.0%

SECONDARY OUTCOMES:
Pathologic complete response rate | post-neoadjuvant chemotherapy; ~ 4-6 months from treatment start
  The rate of pathologic complete response at the primary tumor site from the standard 15% to >20%.

CONTACTS AND LOCATIONS:
Overall Officials: Roshni Rao, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- See also: Related Info — http://www.la-press.com/bootcamp-during-neoadjuvant-chemotherapy-for-breast-cancer-a-randomize-article-a3038